CLINICAL TRIAL: NCT05014295
Title: Patient Recall of Cancer Screening and Diagnosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE1Z21
Record Dates: First submitted 2021-08-13; First posted 2021-08-20 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer; Prostate Cancer
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Survey questions at baseline and at one week. The control group will have had one week to reflect on the questions, and investigators anticipate some influence of this on responses.
- Intervention Group (Active Comparator): The intervention group will be prompted about accessing their medical records from the major local health systems online, with links to directions provided by each hospital system. They will then be asked to fill out the same questionnaire.
  Interventions: Other: Accessing personal medical records online via online portals

INTERVENTIONS:
Other: Accessing personal medical records online via online portals — The participants will receive details on accessing personal medical records online via online portals, for each of the major hospital systems
  Arms: Intervention Group

SUMMARY:
The purpose of this research is to try to better understand how much information relating to cancer screening and diagnoses that people can recall on their own and to better understand how to help people get better information. In this study, investigators will see if giving time or other resources help individuals remember more and more accurate details about their cancer screening and care.

DETAILED DESCRIPTION:
This is a randomized controlled trial of an intervention to encourage use of online medical records for filling out a cancer screening, diagnosis and treatment questionnaire. Participants will be asked to self-report on cancer screening and treatment. They will then be asked the same questions again a week later.

The control group will have had one week to reflect on the questions, and investigators anticipate some influence of this on responses. The intervention group will be prompted about accessing their medical records from the major local health systems online, with links to directions provided by each hospital system. They will then be asked to fill out the same questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with breast or prostate cancer within the last 10 years
* have access to the internet with a working email address
* reside in Northeast Ohio

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-06-22 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Completeness of survey | at 1 week (after second survey completed)
  Completeness: For each survey, for each participant, investigators will count the number of "don't know" response rates. From this, investigators will calculate the percent completeness of the survey.
Accuracy of survey | at 1 week (after second survey completed)
  Investigators will assess the inter-rater reliability between the first and second survey by calculating a Cohen's Kappa coefficient. Although not a perfect assumption, investigators will use the second survey as the reference. Number of changed answers on an individual level will be calculated, representing improved accuracy. Investigators do not anticipate many changes, and, again, this will not be normally distributed.

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Thompson, PhD, Principal Investigator — Case Comprehensive Cancer Center
Locations (1):
- Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No